CLINICAL TRIAL: NCT01614483
Title: Efficacy of Yellow Cassava to Improve Vitamin A Status of Mildly Deficient Primary School Children in Kenya: a Randomized Controlled Trial
Brief Title: Efficacy of Yellow Cassava to Improve Vitamin A Status of Kenyan School Children
Acronym: CASSAVITA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Collaborators: European Commission (Other); University of Nairobi (Other)
Responsible Party: Principal Investigator, Alida Melse, PhD, Wageningen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: INSTAPAWP2YC
Record Dates: First submitted 2012-06-01; First posted 2012-06-08 (Estimated); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Vitamin A Deficiency
Keywords: Vitamin A deficiency; Biofortification; Cassava; B-carotene; School children; Kenya
MeSH Terms: conditions — Vitamin A Deficiency

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Yellow cassava + placebo capsule (Experimental)
  Interventions: Other: Yellow cassava
- White cassava + placebo capsule (Placebo Comparator)
  Interventions: Other: White cassava
- White cassava + B-carotene capsule (Active Comparator)
  Interventions: Other: White cassava

INTERVENTIONS:
Other: Yellow cassava — Daily provision of 375 g boiled yellow cassava for 18 weeks, 6 days/week Daily provision of placebo capsule for 18 weeks, 6 days/week
  Arms: Yellow cassava + placebo capsule
Other: White cassava — Daily provision of 375 g boiled white cassava for 18 weeks, 6 days/ week Daily provision of placebo capsule for 18 weeks, 6 days/ week
  Arms: White cassava + placebo capsule
Other: White cassava — Daily provision of 375 g boiled white cassava for 18 weeks, 6 days/week Daily provision of B-carotene capsule (1400 µg B-carotene)
  Arms: White cassava + B-carotene capsule

SUMMARY:
The overall aim of the project is to provide proof-of-principle that biofortification of cassava with vitamin A is a viable strategy to improve vitamin A status of deficient populations.

DETAILED DESCRIPTION:
Rationale: Vitamin A deficiency is still common in developing countries and has been proven difficult to combat. A promising approach is to replace common crops with varieties that are naturally richer in vitamin A, which is referred to as biofortification. For cassava, yellow β-carotene rich varieties have recently been introduced in Kenya, and these varieties are now ready to be tested for their efficacy to improve vitamin A status in humans.

Objective: The primary objective is to measure the effect of daily consumption of provitamin A biofortified cassava (providing 50% of the age-specific RDA) on vitamin A status in children aged 5-13 years with mild to moderate vitamin A deficiency in Kenya. To determine the bioefficacy of provitamin A carotenoids from biofortified cassava relative to that of a daily B-carotene supplement (comparison with positive control group). Secondary objectives are: 1) to measure the effect of the intervention on immune function indicators and morbidity; 2) to determine to what degree the serum retinol response to the intervention depends on serum concentrations of retinol and zinc at baseline; 3) to determine the effect of the intervention on functional indicators such as dark adaptation capacity, gut integrity, hematology indicators and thyroid status; 4) to determine the mediating effect of SNP's in the BCMO1 gene on treatment outcome.

Study design & Study population : In this randomized controlled trial, school children aged 5-13 years living in the Kibwezi area, Kenya. Children will be selected from three (or four) primary schools in the area that have been pre-selected based on the prevalence of vitamin A deficiency, location and willingness to participate.

Intervention: After screening for eligibility and a 2-week run-in period (n=360) Children will be randomly allocated to three different treatments: 1) 400 g of yellow cassava providing ~50% of the RDA for vitamin A; and a placebo capsule; 2) 400 g of white cassava; and a placebo capsule; 3) 400 g of white cassava and a capsule containing 100 RAE of all-trans β-carotene.

Main study parameters/endpoints: The main outcome measure will be differences in serum retinol concentrations between groups. Other outcome measures include other vitamin A status indicators (β-carotene, retinol binding protein, transthyretin), immune function indicators, dark adaptation, iron status indicators, anthropometrics, gut integrity, and thyroid function.

ELIGIBILITY:
Inclusion Criteria:

* Low vitamin A status (retinol binding protein (RBP) at the lowest end of the distribution will be included in the study)

Exclusion Criteria:

* History or signs of infectious or systemic diseases (e.g. tuberculosis, sickle cell anaemia)
* Anaemia, malaria or acute inflammation at the day of baseline measurements

Ages: 61 Months to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 341 (Actual)
Dates: Start 2012-05; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Change in serum retinol concentration | Baseline, end of study (4 months)

SECONDARY OUTCOMES:
Immune function indicators | End of study (4 months)
  neopterin, IL-2, IL4, IL10, IL13, TNF-a, IFN-γ, TGF-β in serum; IgA in saliva
Bioefficacy | Baseline, end of study (4 months)
  Comparison of change in serum retinol between yellow cassava group and positive control (B-carotene supplement group)
Functional indicators | End of study (4 months)
  Gut integrity, dark adaptation, morbidity
Thyroid function | End of study (4 months
  Serum Tg, TSH
Effect modification | Baseline
  Serum zinc, serum retinol, iron status, polymorphisms
Anemia | End of study (4 months)
  Hemoglobin

CONTACTS AND LOCATIONS:
Overall Officials: Alida Melse, PhD, Principal Investigator — Wageningen University
Locations (1):
- Kibwezi District, Kibwezi, Eastern Kenya, Kenya

REFERENCES:
- [Background] Talsma EF, Brouwer ID, Verhoef H, Mbera GN, Mwangi AM, Demir AY, Maziya-Dixon B, Boy E, Zimmermann MB, Melse-Boonstra A. Biofortified yellow cassava and vitamin A status of Kenyan children: a randomized controlled trial. Am J Clin Nutr. 2016 Jan;103(1):258-67. doi: 10.3945/ajcn.114.100164. Epub 2015 Dec 16. PMID 26675768
- [Background] Talsma EF, Melse-Boonstra A, de Kok BP, Mbera GN, Mwangi AM, Brouwer ID. Biofortified cassava with pro-vitamin A is sensory and culturally acceptable for consumption by primary school children in Kenya. PLoS One. 2013 Aug 30;8(8):e73433. doi: 10.1371/journal.pone.0073433. eCollection 2013. PMID 24023681
- [Background] Talsma EF, Borgonjen-van den Berg KJ, Melse-Boonstra A, Mayer EV, Verhoef H, Demir AY, Ferguson EL, Kok FJ, Brouwer ID. The potential contribution of yellow cassava to dietary nutrient adequacy of primary-school children in Eastern Kenya; the use of linear programming. Public Health Nutr. 2018 Feb;21(2):365-376. doi: 10.1017/S1368980017002506. Epub 2017 Oct 2. PMID 28965533
- See also: Related Info — http://www.instapa.org